CLINICAL TRIAL: NCT00075712
Title: A Randomized Feasibility Trial to Determine the Impact of Timing of Surgery and Chemotherapy in Newly Diagnosed Patients With Advanced Epithelial Ovarian, Primary Peritoneal or Fallopian Tube Carcinoma
Brief Title: Timing of Surgery and Chemotherapy in Treating Patients With Newly Diagnosed Advanced Ovarian Epithelial, Fallopian Tube, or Primary Peritoneal Cavity Cancer
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Royal College of Obstetricians and Gynecologists (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: RCOG-MRC-CHORUS; CDR0000347463 (Registry Identifier: PDQ (Physician Data Query)); EU-20350; ISRCTN74802813
Record Dates: First submitted 2004-01-09; First posted 2004-01-13 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2007-05

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer; Primary Peritoneal Cavity Cancer
Keywords: stage IV ovarian epithelial cancer; stage IIIA fallopian tube cancer; stage IIIB fallopian tube cancer; stage IIIC fallopian tube cancer; stage IV fallopian tube cancer; stage IIIA primary peritoneal cavity cancer; stage IIIB primary peritoneal cavity cancer; stage IIIC primary peritoneal cavity cancer; stage IV primary peritoneal cavity cancer; stage IIIA ovarian epithelial cancer; stage IIIB ovarian epithelial cancer; stage IIIC ovarian epithelial cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Carboplatin; Paclitaxel; Chemotherapy, Adjuvant; Neoadjuvant Therapy

INTERVENTIONS:
Drug: carboplatin
Drug: paclitaxel
Procedure: adjuvant therapy
Procedure: conventional surgery
Procedure: neoadjuvant therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop tumor cells from dividing so they stop growing or die. Giving a chemotherapy drug before surgery may shrink the tumor so that it can be removed; giving chemotherapy after surgery may kill any remaining tumor cells. It is not yet known whether giving chemotherapy before and after surgery is more effective than giving chemotherapy after surgery in treating ovarian epithelial, fallopian tube, or primary peritoneal cavity cancer.

PURPOSE: This randomized phase II/III trial is studying how well giving chemotherapy before and after surgery works and compares it to giving chemotherapy after surgery alone in treating patients with newly diagnosed advanced ovarian epithelial, fallopian tube, or primary peritoneal cavity cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the feasibility of a randomized trial to determine the impact of the timing of surgery and chemotherapy in patients with newly diagnosed advanced ovarian epithelial, primary peritoneal, or fallopian tube cancer.

OUTLINE: This is a randomized, pilot, multicenter study. Patients are randomized to 1 of 2 treatment arms.

* Arm I (primary surgery): Patients undergo radical surgery. Within 6 weeks after primary surgery, patients receive chemotherapy comprising carboplatin alone or in combination with paclitaxel or another chemotherapy agent on day 1. Chemotherapy repeats every 3 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients may undergo interval debulking surgery after the third course of chemotherapy.
* Arm II (neoadjuvant chemotherapy): Patients receive chemotherapy as in arm I for 3 courses. Within 3 weeks after chemotherapy, patients undergo radical surgery. Within 6 weeks after surgery, patients receive an additional 3 courses of chemotherapy as in arm I.

Patients are followed at 9 months after randomization, every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: Approximately 100-150 patients will be accrued for this study within 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Newly diagnosed advanced ovarian epithelial, primary peritoneal, or fallopian tube cancer
* Clinical and imaging evidence of a pelvic mass with extrapelvic metastases within the past 4 weeks
* Serum CA 125/CEA ratio > 25
* Plans to receive carboplatin-based chemotherapy

PATIENT CHARACTERISTICS:

Age

* Adult

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* Considered fit to undergo protocol treatment and follow-up
* No other prior or concurrent malignancy that would preclude study treatment or comparisons

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* See Disease Characteristics

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2003-09

PRIMARY OUTCOMES:
Overall survival at 3 years
Progression-free survival
Quality of life by Quality of Life Questionnaire Core 30 Items (QLQ-C30) and QLQ-ovarian cancer (QLQ-OV28)

CONTACTS AND LOCATIONS:
Overall Officials: Sean Kehoe, Principal Investigator — Oxford University Hospitals NHS Trust
Locations (70):
- United Kingdom (70):
  - Stoke Mandeville Hospital, Aylesbury-Buckinghamshire, England
  - North Devon District Hospital, Barnstaple, England
  - Royal United Hospital, Bath, England
  - Blackpool Victoria Hospital, Blackpool, England
  - Bradford Royal Infirmary, Bradford, England
  - Sussex Cancer Centre at Royal Sussex County Hospital, Brighton, England
  - Broomfield Hospital, Broomfield, England
  - Cumberland Infirmary, Carlisle, England
  - Gloucestershire Oncology Centre at Cheltenham General Hospital, Cheltenham, England
  - Essex County Hospital, Colchester, England
  - Walsgrave Hospital, Coventry, England
  - Derbyshire Royal Infirmary, Derby, England
  - Royal Derby Hospital, Derby, England
  - Birmingham Women's Hospital, Edgbaston, England
  - Royal Devon and Exeter Hospital, Exeter, England
  - Frimley Park Hospital, Frimley, England
  - Queen Elizabeth Hospital, Gateshead, England
  - St. Luke's Cancer Centre at Royal Surrey County Hospital, Guildford, England
  - Hereford Hospitals, Hereford, England
  - Princess Royal Hospital at Hull and East Yorkshire NHS Trust, Hull, England
  - Ipswich Hospital, Ipswich, England
  - Royal Lancaster Infirmary, Lancaster, England
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - Leicester General Hospital, Leicester, England
  - Lincoln County Hospital, Lincoln, England
  - Liverpool Women's Hospital, Liverpool, England
  - Saint Bartholomew's Hospital, London, England
  - Barts and the London School of Medicine, London, England
  - Medical Research Council Clinical Trials Unit, London, England
  - St. George's Hospital, London, England
  - Royal Marsden - London, London, England
  - Hammersmith Hospital, London, England
  - St. Mary's Hospital, Manchester, England
  - Christie Hospital, Manchester, England
  - Wythenshawe Hospital, Manchester, England
  - Clatterbridge Centre for Oncology, Merseyside, England
  - James Cook University Hospital, Middlesbrough, England
  - Milton Keynes General Hospital, Milton Keynes, England
  - Northampton General Hospital, Northampton, England
  - Norfolk and Norwich University Hospital, Norwich, England
  - Oxford Radcliffe Hospital, Oxford, England
  - Derriford Hospital, Plymouth, England
  - Dorset Cancer Centre, Poole Dorset, England
  - Portsmouth Oncology Centre at Saint Mary's Hospital, Portsmouth Hants, England
  - Whiston Hospital, Prescot Merseyside, England
  - Rosemere Cancer Centre at Royal Preston Hospital, Preston, England
  - Oldchurch Hospital, Romford, England
  - Cancer Research Centre at Weston Park Hospital, Sheffield, England
  - Royal Hallamshire Hospital, Sheffield, England
  - Royal Shrewsbury Hospital, Shrewsbury, England
  - Wexham Park Hospital, Slough, Berkshire, England
  - Staffordshire General Hospital, Stafford, England
  - University Hospital of North Staffordshire, Stoke-on-Trent, England
  - St. Peter's Hospital, Surrey, England
  - Great Western Hospital, Swindon, England
  - Taunton and Somerset Hospital, Taunton Somerset, England
  - Torbay Hospital, Torquay, England
  - Walsall Manor Hospital, Walsall, England
  - Good Hope Hospital, West Midlands, England
  - Southend University Hospital NHS Foundation Trust, Westcliff-on-Sea, England
  - Yeovil District Hospital, Yeovil, England
  - Centre for Cancer Research and Cell Biology at Queen's University Belfast, Belfast, Northern Ireland
  - Aberdeen Royal Infirmary, Aberdeen, Scotland
  - Ninewells Hospital, Dundee, Scotland
  - Raigmore Hospital, Inverness, Scotland
  - Ysbyty Gwynedd, Bangor, Wales
  - University Hospital of Wales, Cardiff, Wales
  - Velindre Cancer Center at Velindre Hospital, Cardiff, Wales
  - South West Wales Cancer Institute, Swansea, Wales
  - Wrexham Maelor Hospital, Wrexham, Wales